CLINICAL TRIAL: NCT04856618
Title: Machine Learning-Based Prediction of Major Perioperative Allogeneic Blood Requirements in Cardiac Surgery
Acronym: PREMATRICS
Status: Completed | Type: Observational
Sponsor: Kepler University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PREMATRICS
Record Dates: First submitted 2021-04-16; First posted 2021-04-23 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Transfusion-dependent Anemia
Keywords: Artificial Intelligence; Machine Learning; Transfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Massive Transfusion Positive: Massive Transfusion Positive
  Interventions: Biological: Massive Transfusion of Allogeneic Blood
- Massive Transfusion Negative: Massive Transfusion Negative

INTERVENTIONS:
Biological: Massive Transfusion of Allogeneic Blood — Massive Transfusion of Allogeneic Blood, > pRBCs
  Groups: Massive Transfusion Positive

SUMMARY:
Cardiac surgery is one of the clinical surgical specialties that carries a particularly high risk for patients to suffer from severe bleeding perioperatively and consequent anemia, which subsequently requires transfusion of allogeneic blood.

Although a surprisingly high number of patients in cardiac surgery do not require perioperative transfusions, it is primarily those patients who do require transfusion who are subsequently at risk for a worse outcome.

In recent years many studies have been published discussing measures that can assist physicians in avoiding the triad of anemia, bleeding, and transfusion in cardiac surgery. Within these publications, the implementation of Patient Blood Management (PBM) is advised. PBM is a set of measures aimed at improving patient outcome by reducing perioperative bleeding and thus preventing both anemia and bleeding.

The three pillars of this bundle are the preoperative preparation of anemic patients with iron, erythropoietin, folic acid and vitamin B12, the prevention of intraoperative blood loss and the reasonable indication for allogeneic transfusions.

Nevertheless, it must be mentioned that the implementation of at least part of these measures is laborious, and full implementation of the recommended bundle is therefore rarely achieved. As a consequence, the full potential of Patient Blood Management is not always realized. Unfortunately this means that transfusion of allogeneic blood cannot be prevented in many patients.

A small proportion of patients undergoing cardiac surgery requires a very large amount of allogeneic blood perioperatively. These patients are typically those with a particularly poor outcome. Massive transfusion of allogeneic blood in this situation is an indicator of complications and a cause of increased mortality.

Although cardiac surgeons and anesthesiologists believe they can assess which patients are at high risk for hemorrhage, recent publications indicate that there is an urgent need for adequate predictive methods. A variety of studies exist that attempt to predict perioperative transfusion requirements, but to date have been plagued by several limitations. Either the previous publications do not focus on the prediction of massive transfusion of allogeneic blood, i.e. administration of ten or more packed red blood cell units perioperatively, but on much lower transfusion volumes, have only low predictive strength to predict massive transfusion in daily clinical practice, or are hardly usable for true prediction because they use factors (features) that are not strictly present only in the preoperative phase.

If an accurate prediction model based on a few features could be created and those patients particularly at risk of massive transfusion of allogeneic blood could be identified, it would subsequently be possible to develop an adapted clinical pathway that would allow patient care to be improved and individualized interventions adapted to the situation to be implemented.

In the best case, an adapted care of patients would be possible, which is able to increase the acceptance for the use of even complex measures of patient blood management. This is especially true for measures such as preoperative preparation with iron and/or erythropoietin, the use of a cell saver, and a particularly careful surgical approach.

Even if it is difficult to apply all measures of patient blood management in all patients, it would be possible with an approach as described to identify those patients who would benefit most from individualized approaches.

ELIGIBILITY:
Inclusion Criteria:

* All patients that underwent cardiac surgery at the Kepler University Hospital in the period between 2010-01-01 and 2019-12-31.

Exclusion Criteria:

* Patients below 18 years of age.
* Presence of congenital heart disease.
* Revision surgery of the same patient.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: As described in the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 3782 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
AUROC for Classification of Necessity for Massive Transfusion | 2010-01-01 to 2019-12-31
  AUROC for Classification of Necessity for Massive Transfusion

SECONDARY OUTCOMES:
Confusion Matrix Values | 2010-01-01 to 2019-12-31
  Confusion Matrix Values
Descriptive Statistics | 2010-01-01 to 2019-12-31
  Descriptive Statistics (age, gender, EuroSCORE II, ASA, NYHA, CCS, main surgical procedure, ventricular ejection fraction, endocarditis present, myocardial infarction present, chronic pulmonary disease, immediacy requirement of procedure (elective, emergency), arteriopathy present, diabetes present, previous cardiac surgery done, critical condition present, aortic surgery, pulmonary hypertension present, renal impairment (none, moderate, severe, dialysis)).

CONTACTS AND LOCATIONS:
Locations (1):
- Kepler University Hospital, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tschoellitsch T, Bock C, Mahecic TT, Hofmann A, Meier J. Machine learning-based prediction of massive perioperative allogeneic blood transfusion in cardiac surgery. Eur J Anaesthesiol. 2022 Sep 1;39(9):766-773. doi: 10.1097/EJA.0000000000001721. Epub 2022 Jul 20. PMID 35852544